CLINICAL TRIAL: NCT07151196
Title: The Effect of Smartphone Addiction on Posture, Body Awareness, Physical Activity and Balance in University Students
Brief Title: Impact of Smartphone Addiction on Posture, Body Awareness, Physical Activity, and Balance in University Students
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Istinye University (Other)
Responsible Party: Principal Investigator, HÜSNA GÜZEL, LECTURER, Istinye University
Other Study IDs: istinyeuni
Record Dates: First submitted 2025-08-07; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2024-05

CONDITIONS: Balance Assessment; Postural Instability; Smartphone Addiction
Keywords: balance; smartphone addicition; postural ınstability
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 Smartphone Addiction: Duration of smartphone use, postural disorders, body awareness level, amount of physical activity and balance performance were evaluated in these individuals.
- group 2 non-smartphone addicts: Duration of smartphone use, postural disorders, body awareness level, amount of physical activity and balance performance were evaluated in these individuals.

SUMMARY:
This descriptive cross-sectional study aims to evaluate the effects of smartphone addiction (SA) on posture, body awareness, balance, and physical activity among university students. With the rising popularity of smartphones in recent years, there has been increasing concern about their potential role in postural impairments and balance issues. The study population includes first- and second-year students from the Departments of Dental Services and Therapy-Rehabilitation at Fenerbahçe University School of Health Services.

Smartphone addiction will be assessed using the short form of the Smartphone Addiction Scale; posture will be evaluated using the New York Posture Rating Chart; body awareness will be measured using the Body Awareness Questionnaire (BAQ); balance will be assessed with the Becure Balance System; and physical activity levels will be determined using the International Physical Activity Questionnaire-Short Form (IPAQ-SF).

The study hypothesizes that SA significantly affects these physical and sensory parameters. Based on a power analysis using G*Power, a total sample size of 55 participants was determined. The findings are expected to provide valuable insights into the impact of digital device use on the physical health of young adults.

DETAILED DESCRIPTION:
Over the past decade, smartphones have gained widespread popularity across the globe. A recent study indicated that the prevalence of smartphone addiction (SA) among university students is 26.7% in males and 27.9% in females. The primary distinction between smartphones and earlier mobile phones is that smartphones have full internet access and allow users to easily download any application via modern operating system platforms. Thus, smartphones are increasingly regarded as handheld computers rather than traditional phones Despite the convenience they offer, the pathological use of smartphones has emerged as a new public health concern.

Among the major physical problems associated with excessive internet use-one of the key components of smartphone addiction-are visual disturbances, negative effects of radiation, and postural and skeletal disorders. A study conducted in 2021 demonstrated that smartphone use can lead to significant postural alterations in both sagittal and frontal spinal parameters.

Body awareness refers to an individual's ability to recognize their own body and is a reflection of sensory awareness, encompassing physical, emotional, psychological, and social dimensions. Increasing levels of smartphone addiction have been associated with impaired postural proprioceptive feedback and reduced capacity to maintain proper posture.

Balance is defined as the control of the body's center of gravity and can be described as the dynamic regulation of body posture to prevent falls. No study to date has been found in the literature specifically examining the relationship between smartphone addiction and balance.

Given this context, the current study aims to investigate the impact of smartphone addiction on posture, body awareness, and balance among university students.

ELIGIBILITY:
Inclusion Criteria:

* Being a student of Fenerbahçe University SHMYO Department of Dental Services or Department of Therapy and Rehabilitation
* Volunteering to participate in the study
* Having a smartphone
* Between the ages of 18 and 30

Exclusion Criteria:

- Having a neurological, orthopaedic or metabolic problem or disease that may affect balance, physical activity, posture or body awareness

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals who were students of Fenerbahçe University SHMYO Department of Dental Services or Department of Therapy and Rehabilitation were selected.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
EVALUATION OF SMART PHONE ADDICTION | Day 1
  The participants were administered the Short Form of the Smartphone Addiction Scale (SAS-SF). This scale, developed by Kwon et al., was designed to assess the risk of smartphone addiction among adolescents and consists of 10 items rated on a 6-point Likert scale. The items were scored from 1 to 6, with total scores ranging from 10 to 60. Higher scores indicated a greater risk of addiction. The scale was unidimensional and had no subscales. In the Korean sample, the cutoff scores were 31 for males and 33 for females. In our study, the Turkish version of the scale, whose validity and reliability were established by Noyan et al., was used. Participants were classified as addicted or non-addicted based on the cutoff scores determined by Kwon et al. Additionally, the average daily screen time on participants' phones was recorded.
POSTURE ASSESSMENT | Day 1
  The static postures of the participants were evaluated using the New York Posture Analysis. The New York Posture Analysis assessed postural changes in a total of 13 body regions, including the head, neck, shoulders, back, waist, hips, and ankles, through lateral and posterior observations. Each region was scored as 5 if there was no postural deviation, 3 for moderate deviation, and 1 for severe deviation. The scores from the thirteen regions were summed to obtain a total score ranging from 13 to 65. A total score equal to or greater than 45 was classified as very good; 40-44 as good; 30-39 as moderate; 20-29 as poor; and equal to or less than 19 as bad.
EVALUATION OF BODY AWARENESS | Day 1
  Participants' body awareness was assessed using the Body Awareness Questionnaire (BAQ), originally developed in 1989 by Shields, Mallory, and Simon, and later adapted into Turkish with established validity and reliability. The BAQ is designed to identify whether an individual has a normal or abnormal level of sensitivity to bodily processes. It consists of four subscales-attention to bodily changes and responses, sleep-wake cycle, prediction of illness onset, and prediction of bodily reactions-with a total of 18 items. Participants were asked to rate each item on a scale from 1 to 7 (1 = Not at all true for me, 7 = Completely true for me). The scale is evaluated using the total score, which can range from a minimum of 18 to a maximum of 126. Higher total scores indicated greater body awareness.
BALANCE ASSESSMENT | Day 1
  Static balance was assessed using the Becure Balance System, developed by engineers and physiotherapists as part of a TÜBİTAK project. Based on the WiiFit balance board with custom software, the system evaluated center of pressure distribution and postural sway. The protocol included three conditions: 30 seconds standing with eyes open, 30 seconds standing while using a smartphone (typing the Turkish National Anthem), and 30 seconds standing with eyes closed. Key parameters were changes in center of pressure and postural sway under each condition.
PHYSICAL ACTIVITY ASSESSMENT | Day 1
  International Physical Activity Questionnaire-Short Form (IPAQ-SF):
  The IPAQ-SF scoring involved calculating the time spent walking, performing moderate-intensity, and vigorous-intensity physical activities based on the 7-item questionnaire. Time spent sitting was assessed separately as a single item. The total score was calculated by combining the duration (minutes) and frequency (days) of walking, moderate, and vigorous physical activities.

CONTACTS AND LOCATIONS:
Overall Officials: ELİF SENA DUSGUN, asst. prof., Study Chair — FENERBAHCE UNİVERSİTY; BUSE SERT, PT,PhD (c), Study Chair — MEDİPOL UNİVERSİTY; YELİZ CİRAK, PT,PhD (c), Study Director — FENERBAHCE UNİVERSİTY; HÜSNA GÜZEL, Principal Investigator — FENERBAHCE UNİVERSİTY
Locations (1):
- Fenerbahce University, Istanbul, ATASEHIR, Turkey (Türkiye)